CLINICAL TRIAL: NCT05597254
Title: Facial Skin Clinical and Microbial Profiling From Oral Probiotic Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oriflame Cosmetics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022-00672-01
Record Dates: First submitted 2022-10-11; First posted 2022-10-28 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Healthy; Skin Manifestations
MeSH Terms: conditions — Skin Manifestations | interventions — Probiotics; Niacin; Fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic with niacin and berry extract (Experimental)
  Interventions: Dietary Supplement: Probiotic with niacin and berry extract
- Probiotic without niacin and berry extract (Active Comparator)
  Interventions: Dietary Supplement: Probiotic without niacin and berry extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic with niacin and berry extract — 1 capsule daily of probiotic with niacin supplementation for 8 weeks
  Arms: Probiotic with niacin and berry extract
Dietary Supplement: Probiotic without niacin and berry extract — 1 capsule daily of probiotic without niacin supplementation for 8 weeks
  Arms: Probiotic without niacin and berry extract
Dietary Supplement: Placebo — 1 capsule daily of placebo supplementation for 8 weeks
  Arms: Placebo

SUMMARY:
The goal of this double-blind randomized clinical trial is to investigate the effects on the skin from oral intake of probiotic supplements in healthy adult men and women. The main questions it aims to answer are: • Will probiotic supplementation result in beneficial changes to different skin parameters? • Will probiotic supplementation result in alterations in the skin microbiome? Participants will consume the study product daily for 8 weeks and come in for skin measurements at baseline and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Fully informed with the study specifications.
* Signed consent form prior to commencing the study.
* Motivated for participation in the study, and available over the full test period.
* Healthy skin on the face (i.e., absence of psoriasis, eczemas, erythema, oedema, scars, wounds, lesions, or any other type of inflammatory or autoimmune skin condition).
* Healthy gut (i.e., absence of irritable bowel diseases (IBD), irritable bowel syndrome (IBS), or any other type of inflammatory or autoimmune gut condition).
* No supplementation with probiotic, prebiotic or synbiotic products 2 weeks prior and/or during the whole study period.
* No supplementation with niacin (vitamin B3) 2 weeks prior and/or during the whole study period.
* No significant change in skin care routine (such as injectable cosmetics, skin tanning, etc.) throughout the whole study period.
* No significant change in the diet throughout the whole study period.

Exclusion Criteria:

* Not fulfilling the inclusion criteria.
* Pregnant or lactating 3 months prior to study commencement or during the study.
* Women post menopause.
* Use of antibiotics at least 4 weeks prior and/or during the whole study period.
* Sun-tanned facial skin.
* Participating in another clinical study that could interfere with the present research.
* Presented health problems or specific medications that could adversely affect the study outcome.
* Presented any cutaneous hypersensitivity or allergy to cosmetic products.
* Major surgery on the face one year prior to study commencement.
* Applied any cleansing, topical or moisturizing product (including all make-up products) to the measurement area the morning of assessments at Oriflame Cosmetic AB.
* Exposure to artificial UV light and/or to the sun during the study.
* Special diets (vegan, low carbohydrate, weight loss diet, etc.).
* Significant change in weight one month before or during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Skin Features (pores, wrinkles, colour, pigmentation and redness) at 8 weeks | Day 0, Day 56
  Skin features: Pores, wrinkles, colour, pigmentation and redness
  Site: Cheek, Temple and Forehead - 3 measurement per area. Thus 9 in total.
  Procedure: As per WI091 Standard use of the Miravex Antera 3D Camera V1 and TM089 Skin features measurements Using the Antera 3D V1
  Unit:
  Pores: volume (mm3), index, count, volume/count Wrinkles: overall size, depth (mm), width (mm), Texture: Average Roughness (Ra) Colour variation: DeltaE Pigmentation/redness: average level (concentration per unit area), color variation.
Change from Baseline Skin Features (shininess) at 8 weeks | Day 0, Day 56
  Skin features: Shininess
  Site: Entire face
  Procedure: As per WI044 Standard use of the VISIA-CR2.2 V3 and TM066 Determination Of Skin Brightness Using The Image Pro Plus Shine Macro Test V2
  Unit: Arbitrary unit (AU)
Change from Baseline Skin Features (spot size and color) at 8 weeks | Day 0, Day 56
  Skin features: Spot size and color
  Site: Entire face
  Procedure: As per WI044 Standard use of the VISIA-CR2.2 V3 and TM038 Clinical Determination of Spot Size and Colour
  Unit:
  Color = L*a*b*, Delta E Spot size: volume, count
Change from Baseline Superficial Hydration at 8 weeks | Day 0, Day 56
  Skin feature: Superficial hydration
  Site: Upper cheek - triplicate measurements
  Procedure: As per WI003 Standard use of the Corneometer CM 825 to measure skin moisture V4.
  Unit: Arbitrary unit (AU)
Change from Baseline Skin Barrier Integrity at 8 weeks | Day 0, Day 56
  Skin feature: Skin barrier integrity
  Site: Upper cheek - single measurement
  Procedure: As per WI094 Standard Use of the Delfin Vapometer for Skin Barrier Measurements V1.
  Unit: g/m2h
Change from Baseline Sebum Level at 8 weeks | Day 0, Day 56
  Skin feature: Sebum level
  Site: Forehead - triplicate measurements
  Procedure: As per WI005 Standard use of the Sebumeter SM 815 & MPA 5 to Measure Skin Sebum Levels V2.
  Unit: µg/cm2
Change from Baseline Antioxidant Level at 8 weeks | Day 0, Day 56
  Skin feature: Antioxidant level
  Site: Temple/Cheek area
  Procedure: BioZoom
  Unit: Arbitrary unit (AU)
Change from Baseline Microbial Level at 8 weeks | Day 0, Day 56
  Skin feature: Microbial Level
  Site: Forehead
  Procedure: Damp cotton swab
  Unit: Microbial count by sequencing

SECONDARY OUTCOMES:
Questionnaire on general health and wellbeing | Day 0, Day 28, Day 56
  Subjective measurements of self-rated health aspects using a 9-point hedonic scale (extremely good to extremely bad) at baseline, mid and end of study to access intervention effects

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Lee, Principal Investigator — Global Senior Nutritional Scientist
Locations (1):
- Oriflame Cosmetics, Stockholm, Sweden